CLINICAL TRIAL: NCT05430906
Title: Efficacy and Safety of AK104 (PD-1/CTLA-4 Bispecific Antibody) Combined With Chemotherapy as Neoadjuvant Treatment for Advanced Ovarian Cancer: a Single-arm, Open-label, Multicenter Clinical Study
Brief Title: AK104 Combined With Chemotherapy as Neoadjuvant Treatment for Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-003
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104+chemotherapy (Experimental): Participants received 3-4 neo-adjuvant cycles of AK104 10mg/kg Q3W then [paclitaxel (135-175 mg/m²) or docetaxel (75 mg/m²)] and [carboplatin (AUC5 or 6) or cisplatin (75mg/m²)] Q3W; followed by surgery
  Interventions: Drug: AK104 - Chemotherapy

INTERVENTIONS:
Drug: AK104 - Chemotherapy — AK104 10mg/kg then [paclitaxel (135-175 mg/m²) or docetaxel (75 mg/m²)] and [carboplatin (AUC5 or 6) or cisplatin (75mg/m²)] of each 21-day cycle

SUMMARY:
Previous studies have suggested that immunotherapy combined with chemotherapy as neoadjuvant treatment for ovarian cancer may have a synergistic effect and a manageable safety profile.

AK104 is a bispecific antibody targeting PD-1 and CTLA-4. Therefore, this study aimed to evaluate the efficacy and safety of AK104 combined with chemotherapy as the neoadjuvant treatment for advanced ovarian cancer.

ELIGIBILITY:
Key Inclusion Criteria:

- 1. Woman ≥ 18 and ≤ 75 years old on day of signing informed consent. 2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1. 3. Advanced FIGO stage III to IV patient not able to receive primary debulking surgery for which neo adjuvant chemotherapy is recommended.

4. Have at least one measurable lesion per RECIST 1.1 assessed by investigator. 5. Have adequate organ function.

Key Exclusion Criteria:

* 1. Histological diagnosis of malignant tumor of non-epithelial origin of the ovary, the fallopian tube or peritoneum or borderline tumor of the ovary.

  2. Patients with other active malignancies within 5 years prior to enrollment. 3. Known active autoimmune diseases. 4. Use of immunosuppressive agents within 14 days prior to the first dose of study treatment.

  5. Presence of other uncontrolled serious medical conditions.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Complete(R0) resection rate | Average 4 months after the start of drugs
  The margin of the resected specimen showed no tumour involvement

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At the end of 3-4 cycles of neoadjuvant therapy (each cycle is 21 days)
  The ORR is defined as the percentage of participants having complete response or partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Disease control rate (DCR) | At the end of 3-4 cycles of neoadjuvant therapy (each cycle is 21 days)
  The DCR is defined as the proportion of subjects with complete response, partial response, or stable disease based on RECIST Version 1.1.
Pathological Complete Response (pCR) Rate | One week after the surgery
  The pCR is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
Progression-free survival (PFS) | From the date of the start of drugs to date event, assessed up to 1 years
  Progression-free survival is defined as the time from the start of drugs until the first documentation of disease progression or death due to any cause, whichever occurs first.
Number of participants with adverse events (AEs) | From the first dose of neoadjuvant treatment until 90 days after the last dose of neoadjuvant treatment
Number of participants with surgical complications | Intraoperatively, within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tang, Study Chair — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang C, Dai M, Yang J, Tian W, Huang S, Bi F, Zheng K, Tang J. Patient with HR-proficient advanced ovarian cancer achieved a complete response with Cadonilimab combined chemotherapy (PD-1/CTLA-4 bispecific): a case report and literature review. Gynecol Oncol Rep. 2025 Jun 15;60:101785. doi: 10.1016/j.gore.2025.101785. eCollection 2025 Aug. PMID 40600147